CLINICAL TRIAL: NCT05946499
Title: Correlation Between Vitamin A and E Deficiency With Severity of SARS-COV2 Disease.
Brief Title: Evaluation of Vitamin A and E Deficiency With Severity of SARS-COV-2 Disease: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Balsam Sherif Fahmy, Lecturer, Cairo University
Other Study IDs: Vitamin A and E in COVID-19
Record Dates: First submitted 2023-07-12; First posted 2023-07-14 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: 30 ICU-admitted SARS-CoV-2- infected individuals with ARDS or in need of oxygen supplementation
- Group B: 30 ward-admitted SARS-CoV-2-infected individuals not suffering from ARDS and not in need of oxygen supplementation
- Group C: 30 sex and age-matched normal individuals

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a novel infectious disease that has been spreading worldwide Coronaviridae study group of the International Committee on taxonomy of viruses (2020). The clinical manifestation of COVID-19 can range from asymptomatic infection to critical illness with severe pneumonia, respiratory failure, and death.

Vitamin A is of special interest in the field of infectious diseases, especially for pulmonary infections. It is crucial for the development of normal lung tissue and tissue repair after injury due to infection. Therefore, it may play a role in recovery after severe COVID-19 pneumonia. Vitamin A has immune regulatory functions and positively affects both the innate and adaptive immune cell response.

The anti-oxidant Vitamin E, and trace element selenium, are major components of anti-oxidant defense. Epidemiological studies demonstrate that deficiencies in, either of these nutrients, alters immune responses and viral pathogenicity.

Data concerning vitamin A and E plasma levels in COVID-19 patients are lacking. Therefore, this study aims at characterizing vitamin A and E plasma levels in COVID-19 and analyzing the association of plasma levels with disease severity and outcome.

DETAILED DESCRIPTION:
The aim of the current study is to evaluate the relation of plasma level of Vitamin A and E and their correlation with severity of SARS-COV2 disease.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients by PCR (polymerase chain reaction) test
* Patients aging 18 to 75 years

Exclusion Criteria:

* Patients with known immunodeficiency - Patients with known lung diseases

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID=19 patients recruited from ICU (intensive care Unit) and chest ward
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Correlating between vitamin A and E deficiency and severity of SARS-COV2 | From September 2021 to November 2022
  Evaluation of vitamin A and E deficiency with COVID-19 disease severity

CONTACTS AND LOCATIONS:
Locations (1):
- balsam Sherif Fahmy, Cairo, None Selected, Egypt